CLINICAL TRIAL: NCT07312409
Title: Does Taurine Supplementation Improve Vascular Function and Orthostatic Responses in Long COVID?
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: York University (Other)
Collaborators: Long COVID Web (Unknown); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Heather Edgell, Associate Professor, York University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Edgell Long COVID trial
Record Dates: First submitted 2025-12-17; First posted 2025-12-31 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Long COVID Syndrome
Keywords: Taurine; Vascular; Long COVID; Orthostatic; Cerebrovascular; Heart rate variability
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Intervention Model Description: All participants will receive the same treatment (i.e. taurine supplementation).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Taurine supplementation (Experimental): Participants will take 12-wks of taurine supplementation (2 x 675mg twice daily).
  Interventions: Dietary Supplement: Taurine supplementation

INTERVENTIONS:
Dietary Supplement: Taurine supplementation — Participants will take 12-wks taurine supplementation (2 x 675mg twice daily).

SUMMARY:
Millions have developed Long COVID (LC), and recent findings show an association between taurine deficiency (an amino acid) and symptoms in LC. Cost-effective and accessible interventions are needed to improve welfare and reduce healthcare costs. We will investigate the efficacy of 12-week taurine supplementation, on vascular function and the cardio/cerebrovascular responses to upright posture in LC. We will measure resting vascular function with EndoPAT and ultrasound, resting heart rate variability, and the blood pressure, heart rate, and brain blood flow response to 5 minutes of head-up tilt before and after 12-weeks of taurine supplementation in LC.

DETAILED DESCRIPTION:
Millions of people have been infected by SARS-CoV-2, or COVID-19, and recent estimates suggest that up to 13% have developed Long COVID [1]. The World Health Organization defines Long COVID as "the continuation or development of new symptoms 3 months after the initial SARS-CoV-2 infection, with these symptoms lasting for at least 2 months with no other explanation." SARS-CoV-2 is known to use angiotensin converting enzyme 2 (ACE2) to enter cells [2], and ACE2 is located in endothelial cells throughout the cardiovascular system contributing to significant vascular dysfunction [3]. Indeed, vascular function, as measured by flow-mediated dilation (FMD) has been shown to be impaired in otherwise healthy young COVID-19 survivors just 3-4 weeks after infection [4] and persists for at least 6 months in patients who were hospitalized [5]. Recent work has shown a significant correlation between low plasma taurine levels (a naturally occurring amino acid which can help regulate cardiovascular and inflammation) and Long COVID symptoms, and the recovery of taurine levels was associated with fewer adverse events [6]. Notably, twelve weeks of taurine supplementation has been shown to improve blood pressure and vascular function in pre-hypertension [7]. These improvements could, in turn, improve orthostatic tolerance (i.e. lightheadedness while upright, a common symptom in Long COVID). Thus, the purpose of the current proposal is to investigate the efficacy of 12-wks taurine supplementation on vascular and orthostatic responses in Long COVID. We hypothesize that Long COVID patients will improve their vascular function and orthostatic response after 12-wks of taurine supplementation.

Participants: Drawing on the results of Sun et al. (2016) [7] to calculate a sample size, we used an expected change in FMD of 3.2±4.7% with taurine supplementation, resulting in a sample size of 19. To account for potential participant drop-out, we intend to recruit 30 Long COVID patients aged 18-65, including 15 males and 15 females. As this is a pilot project, we will re-evaluate our sample sizes/statistical power when approximately 8 males and 8 females have been completed [8]. Duration and type of symptoms will be recorded using the Symptom Burden Questionnaire for Long COVID. Autonomic function will be assessed with the COMPASS-31 questionnaire and people with symptoms of orthostatic intolerance and/or vasomotor impairment will be recruited. Sex and gender will be self-identified and used as covariates. Any co-morbidities and medication use will be recorded but not excluded.

Study Design: This will be an interventional open-label single group assignment study. Each lab assessment will take approximately 60 minutes. Participants will come to York University before and after 12-wks taurine supplementation (2 x 675mg twice daily). During the first visit, they will be given the supplements and a Polar heart rate monitor and instructed in its use for home data collection.

1. Vascular function: Resting brachial artery FMD will be measured with Duplex ultrasound imaging according to international guidelines [9]. Briefly, five minutes of forearm vascular occlusion using a blood pressure cuff will be applied while brachial artery diameter and flow are measured before, during and for 3 minutes after cuff occlusion. Peak hyperemic brachial arterial velocity will also be measured using Doppler ultrasound immediately after cuff release. Analysis of FMD will be done with edge-detection software (Quipu) to expedite the analysis and reduce measurement error [10]. Concurrently an EndoPAT device will also be used to measure endothelial function.
2. Orthostatic responses (during supine rest and 5-min 70o head-up tilt): Cardiovascular and respiratory measures: Heart rate will be measured by ECG, blood pressure/cardiac output will be monitored using a beat-by-beat non-invasive blood pressure device (NexFin), brain blood flow will be assessed with transcranial Doppler ultrasound, and respiratory rate will be assessed using a Respitrace. Heart Rate Variability (HRV): HRV provides an indicator of the autonomic control of heart rate (i.e. parasympathetic and sympathetic balance [11]) and will be analyzed using LabChart Pro 8.0 software in the supine and upright postures. Resting HRV will also be assessed using a Polar heart rate device at home, weekly. The heart rate data will be emailed to the students for analysis.

Analysis plan: Each variable described above will be measured before and after the 12-wks taurine supplementation. To test the study hypotheses, repeated measures analysis of variance will be used to examine differences over time (SPSS). Sex, gender, and symptom duration will be covariates.

ELIGIBILITY:
Inclusion Criteria:

* Participants will have had symptoms of Long COVID post-infection for at least 3 months

Exclusion Criteria:

* Inability to undergo tilt table testing for 5 minutes
* Inability to transport selves to York University from their homes
* Inability to speak English, or provide a translator
* Blood clotting disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Orthostatic responses | Baseline and 12-week dietary supplementation.
  Measure cardiovascular and cerebrovascular responses to upright tilt using beat to beat blood pressure, ECG, and transcranial Doppler.
Vascular function | Baseline and 12-week dietary supplementation.
  Flow-mediated dilation and EndoPAT response. These techniques concurrently measure endothelial function using the same protocol.

SECONDARY OUTCOMES:
Heart rate variability | Baseline and 12-week dietary supplementation.
  Variability of resting heart rate will be measured in lab using ECG and at home using a polar heart rate strap.

CONTACTS AND LOCATIONS:
Locations (1):
- York University, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
It is against REB protocol to provide individual data, particularly in small sample size studies.

REFERENCES:
- [Background] Heart rate variability: standards of measurement, physiological interpretation and clinical use. Task Force of the European Society of Cardiology and the North American Society of Pacing and Electrophysiology. Circulation. 1996 Mar 1;93(5):1043-65. No abstract available. PMID 8598068
- [Background] Thijssen DH, Black MA, Pyke KE, Padilla J, Atkinson G, Harris RA, Parker B, Widlansky ME, Tschakovsky ME, Green DJ. Assessment of flow-mediated dilation in humans: a methodological and physiological guideline. Am J Physiol Heart Circ Physiol. 2011 Jan;300(1):H2-12. doi: 10.1152/ajpheart.00471.2010. Epub 2010 Oct 15. PMID 20952670
- [Background] Corretti MC, Anderson TJ, Benjamin EJ, Celermajer D, Charbonneau F, Creager MA, Deanfield J, Drexler H, Gerhard-Herman M, Herrington D, Vallance P, Vita J, Vogel R; International Brachial Artery Reactivity Task Force. Guidelines for the ultrasound assessment of endothelial-dependent flow-mediated vasodilation of the brachial artery: a report of the International Brachial Artery Reactivity Task Force. J Am Coll Cardiol. 2002 Jan 16;39(2):257-65. doi: 10.1016/s0735-1097(01)01746-6. PMID 11788217
- [Background] Wittes J, Brittain E. The role of internal pilot studies in increasing the efficiency of clinical trials. Stat Med. 1990 Jan-Feb;9(1-2):65-71; discussion 71-2. doi: 10.1002/sim.4780090113. PMID 2345839
- [Background] Sun Q, Wang B, Li Y, Sun F, Li P, Xia W, Zhou X, Li Q, Wang X, Chen J, Zeng X, Zhao Z, He H, Liu D, Zhu Z. Taurine Supplementation Lowers Blood Pressure and Improves Vascular Function in Prehypertension: Randomized, Double-Blind, Placebo-Controlled Study. Hypertension. 2016 Mar;67(3):541-9. doi: 10.1161/HYPERTENSIONAHA.115.06624. Epub 2016 Jan 18. PMID 26781281
- [Background] Khoramjoo M, Wang K, Srinivasan K, Gheblawi M, Mandal R, Rousseau S, Wishart D, Prasad V, Richer L, Cheung AM, Oudit GY. Plasma taurine level is linked to symptom burden and clinical outcomes in post-COVID condition. PLoS One. 2024 Jun 5;19(6):e0304522. doi: 10.1371/journal.pone.0304522. eCollection 2024. PMID 38837993
- [Background] Oikonomou E, Souvaliotis N, Lampsas S, Siasos G, Poulakou G, Theofilis P, Papaioannou TG, Haidich AB, Tsaousi G, Ntousopoulos V, Sakka V, Charalambous G, Rapti V, Raftopoulou S, Syrigos K, Tsioufis C, Tousoulis D, Vavuranakis M. Endothelial dysfunction in acute and long standing COVID-19: A prospective cohort study. Vascul Pharmacol. 2022 Jun;144:106975. doi: 10.1016/j.vph.2022.106975. Epub 2022 Mar 3. PMID 35248780
- [Background] Ratchford SM, Stickford JL, Province VM, Stute N, Augenreich MA, Koontz LK, Bobo LK, Stickford ASL. Vascular alterations among young adults with SARS-CoV-2. Am J Physiol Heart Circ Physiol. 2021 Jan 1;320(1):H404-H410. doi: 10.1152/ajpheart.00897.2020. Epub 2020 Dec 11. PMID 33306450
- [Background] Varga Z, Flammer AJ, Steiger P, Haberecker M, Andermatt R, Zinkernagel AS, Mehra MR, Schuepbach RA, Ruschitzka F, Moch H. Endothelial cell infection and endotheliitis in COVID-19. Lancet. 2020 May 2;395(10234):1417-1418. doi: 10.1016/S0140-6736(20)30937-5. Epub 2020 Apr 21. No abstract available. PMID 32325026
- [Background] Hoffmann M, Kleine-Weber H, Schroeder S, Kruger N, Herrler T, Erichsen S, Schiergens TS, Herrler G, Wu NH, Nitsche A, Muller MA, Drosten C, Pohlmann S. SARS-CoV-2 Cell Entry Depends on ACE2 and TMPRSS2 and Is Blocked by a Clinically Proven Protease Inhibitor. Cell. 2020 Apr 16;181(2):271-280.e8. doi: 10.1016/j.cell.2020.02.052. Epub 2020 Mar 5. PMID 32142651
- [Background] Ballering AV, van Zon SKR, Olde Hartman TC, Rosmalen JGM; Lifelines Corona Research Initiative. Persistence of somatic symptoms after COVID-19 in the Netherlands: an observational cohort study. Lancet. 2022 Aug 6;400(10350):452-461. doi: 10.1016/S0140-6736(22)01214-4. PMID 35934007